CLINICAL TRIAL: NCT04454619
Title: Effectiveness of Pre-surgical Hand Washing in Reducing Bacterial Load, Using an Alcoholic Solution of Chlorhexidine Digluconate and Potassium Sorbate
Brief Title: Pre-surgical Antisepsis Using an Alcoholic Solution of Chlorhexidine Digluconate and Potassium Sorbate
Acronym: sorbectol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Ortopedico y Quirurgico del Pie (Other)
Responsible Party: Principal Investigator, Ricardo Becerro de Bengoa Vallejo, Principal Investigator, Centro Ortopedico y Quirurgico del Pie
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RICBEC
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Antisepsis
MeSH Terms: interventions — Solutions; Sorbic Acid

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Crossover design is used
Who Masked: Outcomes Assessor
Masking Description: The samples will be sent to the laboratory with numbers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand antisepsis with propanolol-1 60% (Active Comparator): Effectiveness of pre-surgical hand washing in reducing bacterial load using propanolol-1 60% as control
  Interventions: Drug: Hand antisepsis with Clorhexidine and solution
- Hand antisepsis with Clorhexidina and solution (Experimental): chlorhexidine gluconate with the addition of an alcoholic solution of chlorhexidine digluconate and potassium sorbate.
  Interventions: Drug: Hand antisepsis with Clorhexidine and solution

INTERVENTIONS:
Drug: Hand antisepsis with Clorhexidine and solution — Hand antisepsis by scrub Surgical Hand scrubbing using chlorhexidine digluconate with the addition of an alcoholic solution of chlorhexidine digluconate and potassium sorbate. both hands using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side
  Other Names: Clorhexidine and alholic solution dicluconate cloehexidine and potassium sorbate

SUMMARY:
The present study evaluates the effects of bactericidal load reduction after surgical hand scrub antisepsis using the reference antiseptic product propan-ol-1 60% as control versus a surgical hand scrub antisepsis with addition of a solution of chlorhexidine digluconate and potassium sorbate in order to test if pass the standard european norm 12791.

DETAILED DESCRIPTION:
The investigators conducted a crossover clinical trial to evaluate the antiseptic effectiveness of preoperative surgical scrubbing using propan-ol-1 60% by scrub using the reference antiseptic product propan-ol-1 60% as control versus a surgical hand scrub antisepsis with addition of a solution of chlorhexidine digluconate and potassium sorbate in order to test if pass the standard european norm 12791. Samples will be taken from the hands of each volunteer after a surgical hands antiseptic.

ELIGIBILITY:
Inclusion Criteria:

* Participants without systemic pathologies, with healthy skin of the hands and short fingernails.
* They do not use substances with antibacterial action.

Exclusion Criteria:

* Taken antibiotics before 10 days of the intervention.
* Wear any jewellery on the hands

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2020-07-18 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Change of bacterial load measured in CFU immediately after hand scrub | Change from bacterial load at 5 minutes
  Participants will scrub the antiseptic solution vigorously from hand to the wrists according with the standard handrub procedure

SECONDARY OUTCOMES:
Change of bacterial loadmeaured in CFU after 3 hours of hand scrub | Change from bacterial load at 3 hours
  Participants will scrub the antiseptic solution vigorously from hand to the wrists according with the standard handrub procedure after 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Becerro de Bengoa Vallejo, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Centro ortopedico y quirurgico del pie, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
A number will be assigned to each participant